CLINICAL TRIAL: NCT03961607
Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Moderate or Severe Acne#a Randomized, Open-label Trial
Brief Title: Conventional Photodynamic Therapy vs. Painless Photodynamic Therapy for Moderate or Severe Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Director, Clinical Professor, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-10
Record Dates: First submitted 2019-05-19; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Acne
Keywords: Photodynamic Therapy; Conventional; Painless; Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluator assesses photographs without prior knowledge of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painless Photodynamic Therapy(P-PDT) group (Experimental): The painless photodynamic therapy group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 150 J/cm2) after applying 5% 5-aminolevulinic acid#ALA#cream for 30min. A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy
- Conventional Photodynamic Therapy(C-PDT) group (Active Comparator): The conventional photodynamic therapy(C-PDT) group underwent narrow-band light-emitting diode (LED) irradiation (630 nm; 50 J/cm2) after applying 5% 5-aminolevulinic acid cream for 1.5h.A repeat treatment was administered once weekly for a maximum of 3 weeks.
  Interventions: Procedure: Aminolevulinic acid photodynamic therapy

INTERVENTIONS:
Procedure: Aminolevulinic acid photodynamic therapy — Aminolevulinic acid photodynamic therapy

SUMMARY:
This study is being done to compare a new, continuous illumination and short Incubation time regimen of aminolevulinic acid photodynamic therapy#ALA- PDT) to a conventional regimen for treatment of Moderate or Severe Acne. The hypothesis is that the continuous illumination approach will be less or even no painful, but equally efficacious, as the old regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed with moderate to severe acne;
2. Male and female patients of age between 18-30 years old ;
3. All patients read the instructions of the subject, willing to follow the program requirements;
4. No other topical treatment received within 2 weeks prior to enrollment;
5. No systemic treatment was given within 4 weeks prior to enrollment;
6. Patients were unsuitable for surgery for various reasons,unwilling to undergo surgery, and signed informed consent when they had informed other alternatives and agreed to take pictures of the lesion. -

Exclusion Criteria:

1. Those who did not complete the informed consent;
2. The lesions belongs to any of the following conditions: There is damage and inflammation, which may lead to the drug entering the open wound;
3. Patients with skin photoallergic diseases, porphyria;
4. Known to have a history of allergies to test drugs (porphyrins) and their chemically similar drugs;
5. Patients with other obvious diseases that may affect the evaluation of efficacy;
6. Scars or patients with a tendency to form scars;
7. Known to have severe immune dysfunction, or long-term use of glucocorticoids and immunosuppressants;
8. Severe heart, liver, kidney disease; with hereditary or acquired People with sexual coagulopathy;
9. Those with severe neurological, psychiatric or endocrine diseases; (10)Women who are pregnant, breast-feeding or using inappropriate contraceptives; those with a history of drug abuse; those who have participated in other drug clinical trials within 4 weeks before treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Moderate or Severe Acne | The clearance rate of Moderate or Severe Acne will be measured at one month after the last treatment
  The clearance rate of Moderate or Severe Acne will be measured at one month after the last treatment

SECONDARY OUTCOMES:
Pain assessment | Immediately, 1st minute, 3rd minute, 5th minute, 7th minute, 10th minute and 2 hours, 12 hours, 24hours and 48 hours after treatment
  The pain will be assessed using Visual Analogue Scale#VAS) with a score range of 0-10. The higher the score, the greater the pain, with 0 being no pain and 10 being the most unbearable pain. Pain will be measured at different time points during and after every treatment #including immediately, 1st min, 3rd min, 5th min, 7th min, 10th min and 2nd h, 12th h, 24th h and 48th h after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, PhD, MD, Study Chair — Shanghai Skin Disease Hospital
Locations (1):
- Yunfeng Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed